CLINICAL TRIAL: NCT02422004
Title: Healing of Human Achilles Tendon Rupture: Loading Pattern After Surgical Repair to Achieve Optimal Mechanical Properties and Clinical Outcome
Brief Title: Healing of Human Achilles Tendon Rupture
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bispebjerg Hospital (Other)
Collaborators: University of Copenhagen (Other); Danish Council for Independent Research (Other)
Responsible Party: Principal Investigator, Pernilla Eliasson, Postdoc, Bispebjerg Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BBH100
Record Dates: First submitted 2015-04-16; First posted 2015-04-21 (Estimated); Last update posted 2015-04-21 (Estimated); Status verified 2015-04

CONDITIONS: Achilles Tendon Rupture
Keywords: Rehabilitation; Weight-bearing; Range of motion
MeSH Terms: interventions — Range of Motion, Articular

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Control (Active Comparator): This constitutes the currently accepted regime and is therefore consider the control group (CTRL) with early range of motion and early weight bearing. The control group was allowed to have partial weight-bearing from day 0 and full weight-bearing from week 4. Furthermore, they were instructed in tendon strain exercise identical with the range of motion group.
  Interventions: Other: Range of motion
- Range of motion (Experimental): Early range of motion and delayed weight bearing (ROM). The range of motion group was restricted completely from weight-bearing until week 6, allowed partial weight-bearing after 6 weeks and full weight-bearing after 8 weeks. In addition to this, the patients were instructed to perform tendon strain exercises, five times a day, from week 2. The exercises were performed by removing the foot from the brace and then perform light dorsal ankle movement, 25 repetitions/time, when sitting on a table.
  Interventions: Other: Range of motion; Other: Delayed weight-bearing
- Immobilization (Experimental): Delayed weight-bearing or range of motion (IMMOB). The immobilization group was restricted completely from weight-bearing until week 6, allowed partial weight-bearing after 6 weeks and full weight-bearing after 8 weeks.
  Interventions: Other: Delayed weight-bearing

INTERVENTIONS:
Other: Range of motion — 25 range of motion exercises of the ankle, 5 times per day.
  Arms: Control; Range of motion
Other: Delayed weight-bearing — No weight-bearing during the first six weeks, and partial weight-bearing during the two following weeks
  Arms: Immobilization; Range of motion

SUMMARY:
The overall aim of this project is to investigate the healing processes of human tendon after suturing a ruptured Achilles tendon, and more specifically to determine the optimal loading pattern of the tendon during the rehabilitation period to ensure complete and good recovery of tendon structure and function. The investigators hypothesize that restricting early weight bearing and only allowing for passive stretching in the early phase of tendon healing will ensure better tissue regeneration and thereby prevent chronic tendon elongation and improve tendon tissue recovery and the clinical outcome.

DETAILED DESCRIPTION:
Surgical repair of Achilles tendon ruptures is known to significantly reduce the risk of re-rupture and to accelerate the time to return to activity compared with non-surgical treatments (1, 2). Although sutured, Achilles tendon rupture requires an extended rehabilitation period following surgery to function normally again. However, the currently available information on this post-operative treatment suggest that the currently available rehabilitation guidelines, which includes early weight bearing, does not accomplish optimal recovery of muscle-tendon function. It has been demonstrated that reduced capacity to perform heel-rises, diminished range of motion of the ankle joint, and reduced calf muscle mass is correlated with a delay in return to activity, and all of these factors could be related to elongation of the healing tendon (3). Importantly, it appears that preventing tendon elongation during rehabilitation improves the clinical outcome, but the actual mechanism for the elongation and thus how to prevent it remains unknown (4). With newly developed techniques in our laboratory we will determine the mechanical properties of human whole Achilles tendon, in vivo, which makes it possible to explore how tendons respond to the regimes following a suture repair and rehabilitation regime.

In contrast to the current rehabilitation regime after tendon surgery, which includes early high loading (weight bearing) already in the first weeks after surgery, we hypothesize that avoiding early weight bearing but allowing for early passive ankle joint range of motion (tissue strain with minimal loading) will prevent chronic tendon elongation, increase tendon stiffness, increase calf strength and muscle volume/thickness, and thus improve the long-term clinical outcome after tendon rupture in humans.

Patients with acute Achilles tendon ruptures will undergo a standardized suture repair (a.m. Kessler) using resorbable suture (Vicryl size 1) at Bispebjerg Hospital and be placed in a brace that inhibits ankle joint movement. During surgery, patients will get four tantalum beads with a diameter of 1.0 mm implanted with a venflon needle in the proximal and the distal stub of the tendon. Thereafter they will be randomized to three post-operative treatment regimes:

Control, range of motion or immobilized

From the currently available data (4, 5, 6) it is suggested that the brace is worn for 6 weeks after surgery in all three groups of the present experiment. The control group will be allowed partial weight-bearing from day 0 and full weight-bearing from week 4, toe rises after 16 weeks, jogging after 24 weeks and return to sports 34 weeks after. The two delayed weight-bearing groups (range motion group and immobilized group) will be restricted completely from weight-bearing initially (6 weeks), allowed partial weight-bearing after 6 weeks and full weight-bearing after 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Complete Achilles tendon rupture placed in the mid-substance of the Achilles tendon
* Presented within 14 days from injury

Exclusion Criteria:

* re-rupture
* other injuries affecting their lower limb functions
* systemic diseases influencing tendon healing
* immunosuppressive treatment including systemic corticosteroid treatment
* inability to follow rehabilitation or follow-ups.

Ages: 18 Years to 67 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2012-08; Primary Completion 2016-09 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
Tendon elongation | 2, 6, 12, 26 and 52 weeks after rupture
  Tendon elongation will be evaluated using x-ray and measurements of the distance between tantalum beads

SECONDARY OUTCOMES:
Heel-rise | 26 and 52 weeks after rupture
  The number of heel-rises and the heel-rise height will be used for
  calculation of the heel-rise work.
Achilles tendon total rupture score (ATRS) | 12, 26 and 52 weeks after rupture
  Patient reported outcome regarding function in their Achilles tendon
Elastic modulus of the tendon | 6, 26 and 52 weeks after rupture
  Tendon stiffness will be evaluated during a voluntary plantar flexion contraction where force and tendon elongation is measured using a force transducer and x-ray, respectively. Tendon size will be evaluated by MRI. Elastic modulus will be calculated based on stiffness and size of the tendon.
Range of motion test | 26 and 52 weeks after rupture
  Range of motion in the ankle will be measured.
Victorian Institute of Sport Assessment questionnaire - Achilles tendinopathy (VISA-A) | 12, 26 and 52 weeks after rupture
  Patient reported outcome regarding pain in their Achilles tendon.
Plantar flexion muscle strength | 26 and 52 weeks after rupture
  Plantar flexion muscle strength will be measured during a maximal voluntary isometric contraction with ankle flexion at -10, 0˚ of dorsiflexion
Calf muscle size | 6, 26 and 52 weeks after rupture
  Calf muscle size will be assessed using MRI.
Tendon size | 6, 26 and 52 weeks after rupture
  Tendon size will be assessed using MRI.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Magnusson, PT, DSc, PhD, Study Director — Bispebjerg Hospital, University of Copenhagen; Michael Kjaer, MD, PhD, Study Director — Bispebjerg Hospital, University of Copenhagen
Locations (1):
- Bispebjerg Hospital, Copenhagen, Denmark

REFERENCES:
- [Background] Magnusson SP, Narici MV, Maganaris CN, Kjaer M. Human tendon behaviour and adaptation, in vivo. J Physiol. 2008 Jan 1;586(1):71-81. doi: 10.1113/jphysiol.2007.139105. Epub 2007 Sep 13. PMID 17855761
- [Background] Maffulli N, Waterston SW, Squair J, Reaper J, Douglas AS. Changing incidence of Achilles tendon rupture in Scotland: a 15-year study. Clin J Sport Med. 1999 Jul;9(3):157-60. doi: 10.1097/00042752-199907000-00007. PMID 10512344
- [Background] Saxena A, Ewen B, Maffulli N. Rehabilitation of the operated achilles tendon: parameters for predicting return to activity. J Foot Ankle Surg. 2011 Jan-Feb;50(1):37-40. doi: 10.1053/j.jfas.2010.10.008. Epub 2010 Nov 24. PMID 21106412
- [Background] Andersson T, Eliasson P, Aspenberg P. Tissue memory in healing tendons: short loading episodes stimulate healing. J Appl Physiol (1985). 2009 Aug;107(2):417-21. doi: 10.1152/japplphysiol.00414.2009. Epub 2009 Jun 18. PMID 19541735
- [Background] Mortensen HM, Skov O, Jensen PE. Early motion of the ankle after operative treatment of a rupture of the Achilles tendon. A prospective, randomized clinical and radiographic study. J Bone Joint Surg Am. 1999 Jul;81(7):983-90. doi: 10.2106/00004623-199907000-00011. PMID 10428130
- [Background] Kangas J, Pajala A, Ohtonen P, Leppilahti J. Achilles tendon elongation after rupture repair: a randomized comparison of 2 postoperative regimens. Am J Sports Med. 2007 Jan;35(1):59-64. doi: 10.1177/0363546506293255. Epub 2006 Sep 14. PMID 16973901
- [Derived] Eliasson P, Agergaard AS, Couppe C, Svensson R, Hoeffner R, Warming S, Warming N, Holm C, Jensen MH, Krogsgaard M, Kjaer M, Magnusson SP. The Ruptured Achilles Tendon Elongates for 6 Months After Surgical Repair Regardless of Early or Late Weightbearing in Combination With Ankle Mobilization: A Randomized Clinical Trial. Am J Sports Med. 2018 Aug;46(10):2492-2502. doi: 10.1177/0363546518781826. Epub 2018 Jul 2. PMID 29965789